CLINICAL TRIAL: NCT02214628
Title: A 24 Month Phase 2A Open Label Safety Study of Fovista® (Anti-PDGF-BB Pegylated Aptamer) Regiment Administered in Combination With Avastin®, Eylea®, or Lucentis®) During the Induction and Maintenance Phase of Therapy
Brief Title: Phase 2A Open Label Safety Study of Fovista® (Anti-PDGF BB) Regimen Administered in Combination With Anti-VEGF Therapy to Study Sub-Retinal Fibrosis in Neovascular AMD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Ophthotech Corporation (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPH1005
Record Dates: First submitted 2014-08-05; First posted 2014-08-12 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2019-01

CONDITIONS: Age-related Macular Degeneration
Keywords: Wet AMD; Choroidal neovascularization; Fovista®; E10030; Avastin®; Eylea®
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fovista® plus anti-VEGF Simultaneous (Experimental): Subjects will be administered Fovista® (anti-PDGF BB) plus anti-VEGF as a "Simultaneous" regimen followed by quarterly administration.
  Interventions: Drug: Fovista® (anti-PDGF BB) plus anti-VEGF
- Fovista® plus anti-VEGF Pre-Treatment (Experimental): Subjects will be administered Fovista® (anti-PDGF BB) plus anti-VEGF as a "Pre-Treatment" regimen followed by quarterly administration.
  Interventions: Drug: Fovista® (anti-PDGF BB) plus anti-VEGF

INTERVENTIONS:
Drug: Fovista® (anti-PDGF BB) plus anti-VEGF
  Other Names: Fovista®; anti-VEGF

SUMMARY:
The objective is to evaluate the safety of intravitreal Fovista® (anti-PDGF BB) administered in combination with anti-VEGF therapy.

DETAILED DESCRIPTION:
The objective is to evaluate the safety of intravitreal Fovista® (anti-PDGF BB) administered in combination with anti-VEGF therapy in either a "Simultaneous" Regimen (Fovista® administered with anti-VEGF same day) or "Pre-Treatment" Regimen (monotherapy Fovista® Day 0 followed by Fovista® administered in combination with anti-VEGF Day 2).

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender aged ≥ 50 years
* All fluorescein angiographic subtypes with presence of active choroidal neovascularization

Exclusion Criteria:

* Any intraocular surgery or thermal laser within three (3) months of trial entry. Any prior thermal laser in the macular region, regardless of indication
* Subjects with subfoveal scar or subfoveal atrophy
* Any ocular or periocular infection in the past twelve (12) weeks
* History of any of the following conditions or procedures in the study eye: Rhegmatogenous retinal detachment, pars plana vitrectomy, filtering surgery (e.g. trabeculectomy), glaucoma drainage device, corneal transplant

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Phoenix, Arizona
  - Beverly Hills, California
  - Sacramento, California
  - Santa Ana, California
  - Augusta, Georgia
  - Oak Forest, Illinois
  - Boston, Massachusetts
  - Jackson, Michigan
  - Minneapolis, Minnesota
  - Cincinnati, Ohio
  - Ladson, South Carolina
  - Abilene, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Fovista® (Anti-PDGF BB) Plus Anti-VEGF Simultaneous Regimen: Subjects administered Fovista® (anti-PDGF BB) plus anti-VEGF as a "Simultaneous" regimen followed by quarterly administration.
- Fovista® (Anti-PDGF BB) Plus Anti-VEGF Pre-Treatment Regimen: Subjects administered Fovista® (anti-PDGF BB) plus anti-VEGF as a "Pre-Treatment" regimen followed by quarterly administration
Period: Overall Study
Arm/Group | Fovista® (Anti-PDGF BB) Plus Anti-VEGF Simultaneous Regimen | Fovista® (Anti-PDGF BB) Plus Anti-VEGF Pre-Treatment Regimen
Started | 63 | 38
Completed | 36 | 9
Not Completed | 27 | 29

BASELINE CHARACTERISTICS:
Groups:
- Fovista® (Anti-PDGF BB) Plus Anti-VEGF Simultaneous: Subjects administered Fovista® (anti-PDGF BB) plus anti-VEGF as a "Simultaneous" regimen followed by quarterly administration
- Total: Total of all reporting groups
Arm/Group | Fovista® (Anti-PDGF BB) Plus Anti-VEGF Simultaneous | Fovista® (Anti-PDGF BB) Plus Anti-VEGF Pre-Treatment Regimen | Total
Number analyzed (Participants) | 63 | 38 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 9
  >=65 years | 60 | 32 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.3 (7.92) | 74.8 (9.89) | 77.0 (8.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 29 | 69
  Male | 23 | 9 | 32
Region of Enrollment [Number; unit: participants]
  United States | 63 | 38 | 101

OUTCOME MEASURES:

1. Primary Outcome: Number of Subject With Non Serious Adverse Events (Reported by >5% of Subjects)
Description: Number of subjects on either arm with non-serious adverse events (reported by >5% of subjects)
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Fovista® (Anti-PDGF BB) Plus Anti-VEGF Simultaneous Regimen | Fovista® (Anti-PDGF BB) Plus Anti-VEGF Pre-Treatment Regimen
Number analyzed (Participants) | 63 | 38
Participants | 51 | 34

2. Primary Outcome: Number of Subjects With Serious Adverse Events
Description: Number of subjects with serious adverse events in each arm
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Fovista® (Anti-PDGF BB) Plus Anti-VEGF Simultaneous Regimen | Fovista® (Anti-PDGF BB) Plus Anti-VEGF Pre-Treatment Regimen
Number analyzed (Participants) | 63 | 38
Participants | 19 | 8

ADVERSE EVENTS:
Time Frame: Up to a maximum exposure of 24 months
Arm/Group | Fovista® (Anti-PDGF BB) Plus Anti-VEGF Simultaneous Regimen | Fovista® (Anti-PDGF BB) Plus Anti-VEGF Pre-Treatment Regimen
All-Cause Mortality (participants affected / at risk) | 2/63 | 2/38
Serious Adverse Events (participants affected / at risk) | 19/63 | 8/38
Other Adverse Events (participants affected / at risk) | 51/63 | 34/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fovista® (Anti-PDGF BB) Plus Anti-VEGF Simultaneous Regimen (N=63) | Fovista® (Anti-PDGF BB) Plus Anti-VEGF Pre-Treatment Regimen (N=38)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Surgical failure (General disorders) | 1 (1) | 0 (0)
Biloma (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Appendiceal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Endophthalmitis (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (2) | 0 (0)
Facial bone fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (5) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Perirenal haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastasis to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Ischemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fovista® (Anti-PDGF BB) Plus Anti-VEGF Simultaneous Regimen (N=63) | Fovista® (Anti-PDGF BB) Plus Anti-VEGF Pre-Treatment Regimen (N=38)
Nasopharyngitis (Infections and infestations) | 8 (10) | 4 (4)
Sinusitis (Infections and infestations) | 7 (7) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (7) | 3 (3)
Cataract (Eye disorders) | 6 (9) | 2 (6)
Conjuctival haemorrhage (Eye disorders) | 31 (87) | 20 (42)
Eye Pain (Eye disorders) | 9 (11) | 3 (6)
Intraocular pressure increased (Eye disorders) | 9 (12) | 9 (26)
Neovascular age-related macular degeneration (Eye disorders) | 13 (13) | 3 (3)
Retinal haemorrhage (Eye disorders) | 5 (10) | 1 (1)
Visual acuity reduced (Eye disorders) | 2 (2) | 3 (3)
Vitreous detachment (Eye disorders) | 7 (7) | 1 (1)
Vitreous floaters (Eye disorders) | 4 (6) | 3 (3)
Lacrimation increased (Eye disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution agrees not to individually publish the results of the Study without Ophthotech's prior written consent. Institution may participate in a joint, multi-center publication of the Study results with other investigators and/or institutions only, upon the prior written consent of Ophthotech.